CLINICAL TRIAL: NCT03831165
Title: Effects of Melatonin in the Treatment of Genital Herpes
Brief Title: Melatonin Effects on Genital Herpes in Brazilian Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1215208
Record Dates: First submitted 2018-07-03; First posted 2019-02-05 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2020-01

CONDITIONS: Genital Herpes
Keywords: acyclovir; melatonin
MeSH Terms: conditions — Herpes Genitalis | interventions — Melatonin; Acyclovir

STUDY DESIGN:
Intervention Model Description: The patients will be divided into three groups. One group (group A) will receive a bottle with 360 pills of acyclovir 200 mg. These individuals will be instructed to take 2 tablets of 200mg acyclovir (400 mg) twice daily for 90 days. Group B will receive 90 tablets of 30 mg of melatonin, the tablet will be used as 01 tablet daily for 90 days. Group C will receive 90 tablets of melatonin 3mg, and 360 tablets of acyclovir dose is 1 tablet per day for 90 days.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patients will be treated at the Clinic of Gynecology, University of Sao Paulo during a total of 04 visits. In the first and fourth visits, patients will be sent to the laboratory of the University Hospital for collecting the cluster of differentiation 4 cells, interleukin-2 and serology for herpes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- melatonin 3mg + Acyclovir 400mg (Experimental): Group I - melatonin 3mg + Acyclovir 400mg
  Interventions: Combination Product: Melatonin 3 mg; Drug: Acyclovir
- Acyclovir 400mg (Active Comparator): Group II - Acyclovir 400mg twice a day
  Interventions: Combination Product: Melatonin 3 mg; Drug: Acyclovir
- placebo + melatonin 3mg (Placebo Comparator): Group III - placebo + melatonin 3mg
  Interventions: Combination Product: Melatonin 3 mg; Drug: Acyclovir

INTERVENTIONS:
Combination Product: Melatonin 3 mg — melatonin and placebo
Drug: Acyclovir — Only acyclovir 200 mg twice a day

SUMMARY:
Genital herpes is a common and increasingly-common infection worldwide. The annual incidence in the United States is 1.75 per 1000 inhabitants. The etiologic agent is the herpes type 1 and 2 strains simplex virus. Classical Treatment is with acyclovir which decreases the duration of the disease and prevents rashes but has no curative effect. Also, studies show herpes resistance to acyclovir which has stimulating research into new drugs to treat this condition. Authors suggest melatonin way be a therapeutic agent in herpetic disease due to its modulatory action in immune and inflammatory responses when administered in adequate doses. Therefore, the aim of this study is to evaluate the effects of melatonin in the treatment of genital herpes as well as compare it to acyclovir in a double-blind, prospective and randomized, investigation. Outcome measures will include clinical evaluation of patients and laboratory endpoints.

DETAILED DESCRIPTION:
The authors have investigate the relationship of estrogen-dependent malignant tumors with reduced levels of melatonin. It is speculated that the indoleamine can be classified as anti-estrogenic drug, both by its action on estrogen synthesis with aromatase inhibition and by its interference with estrogen receptors. Experimentally melatonin prevents promotion and growth of mammary tumors in rodents, probably by interacting with epithelial cell receptor; increasing local immunity by acting as an antioxidant agent and by inhibiting telomerase activity in tumor cells .

ELIGIBILITY:
Inclusion criteria:

* clinical and laboratory diagnosis of genital herpes
* real time polymerase chain reaction for herpes type 2
* serology

Exclusion criteria:

* immunodeficiencies
* pregnant women

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female only
Enrollment: 90 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Clinical disease activity | 2 years
  Number of participants with clinical signals of herpes genial activity

CONTACTS AND LOCATIONS:
Overall Officials: Edmund C Baracat, PhD, Study Director — Universidade de Sao Paulo General Hospital
Locations (2):
- Brazil (2):
  - Avenida Doutor Eneas Carvalho de Aguiar 255 10 andar, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No